CLINICAL TRIAL: NCT05547802
Title: Evaluation of the Efficacy of BBIBP-CorV Inactivated Vaccine Combined With BNT62b2 mRNA Booster Vaccine
Brief Title: Serology After BBIBP-CorV Inactivated Vaccine Combined With BNT62b2 mRNA Booster Vaccine
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Béla Nagy Jr., MD, PhD, associate professor, University of Debrecen
Other Study IDs: UDebrecen
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Basic BBIBP-CorV Vaccination is Not as Effective as BNT162b

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples were stored prior to laboratory analysis by an immunoassay to measure the level of anti-SARS-CoV-2 total Ig.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heterologous vaccination cohort: Subjects with two doses of BBIBP-CorV vaccine and third (second booster) dose of the BNT162b2 vaccine.
  Interventions: Biological: BBIBP-CorV and/or BNT162b2 vaccine
- Homologous vaccination cohort: Subjects receiving three doses of BNT162b2 vaccine.
  Interventions: Biological: BBIBP-CorV and/or BNT162b2 vaccine

INTERVENTIONS:
Biological: BBIBP-CorV and/or BNT162b2 vaccine — Booster immunization was carried out at least 4 months after the first two doses of basic immunization.

SUMMARY:
In this prospective study, SARS-CoV-2 spike protein specific total immunoglobulin (Ig) levels are analyzed before and after BNT162b2 third mRNA booster vaccination in individuals previously administered with two doses of BBIBP-CorV vaccine in comparison to immunized participants with three doses of BNT162b2 vaccination. Questionnaires from recruited participants are reviewed prior to booster vaccination for the occurrence of a previous SARS-CoV-2 infection and hospitalization.

DETAILED DESCRIPTION:
Sixty-one volunteers (39 females, 22 males) vaccinated by BBIBP-CorV were included with the mean age of 63.9 years. To serve as a control group, 61 patients (41 females, 20 males) were vaccinated with BNT162b2 at a mean age of 59.9 years. At least four months after the first two-dose vaccination regimens, both groups received the third booster BNT162b2 vaccine based on the recommendations of the Hungarian Public Health Centre. Total Ig levels against SARS-CoV-2 spike protein 1 receptor-binding domain (anti-SARS-CoV-2 S1-RBD) were measured by an immunoassay (Roche Diagnostics) and their calculated ratios after/before booster dose were compared between the two groups. Vaccination efficacy via incidence of infection and hospitalization was monitored during study period. We found that BNT162b2 can successfully booster the effect of two-dose BBIBP-CorV vaccination to enhance humoral immune response against SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria: -

Exclusion Criteria: included age < 18 years, known primary immunodeficiency, malignancy and ongoing immunosuppressive therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of the regular clinical practice, all participants received the third vaccine dose at a general practitioner's (GP) office. Following the initial immunization period, a survey was conducted to monitor vaccine efficacy via the incidence of infection and hospitalization by patient questionnaire. Booster immunization was carried out at least 4 months after the first two doses of basic immunization (two doses of BNT162b2 or BBIBP-CorV), and baseline (pre-booster) antibody level was measured on the same day of the administration of booster immunization (first sampling). Following the booster dose with BNT162b2, another serum sample was collected after 30 days in order to determine induced total level of anti-SARS-CoV-2 spike protein antibodies (second sampling).
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Serology status after booster vaccination | 30 days
  Following the booster dose, serum sample was collected after 30 days to determine induced total level of anti-SARS-CoV-2 spike protein antibodies.

SECONDARY OUTCOMES:
Development of COVID-19 disease | Half year
  Vaccination efficacy via incidence of infection and hospitalization was monitored during study period.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Szekanecz, MD, PhD, Study Director — University of Debrecen
Locations (1):
- University of Debrecen, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: No
These data will be published in a manuscript in a peer-reviewed international journal.